CLINICAL TRIAL: NCT02260258
Title: Neuromuscular Blockade for Post-Cardiac Arrest Care
Acronym: NMB_in_CA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Brigham and Women's Hospital (Other); University of Alabama at Birmingham (Other); Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Michael Donnino, Michael Donnino MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014P000204; 14GRNT20010002 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2014-09-24; First posted 2014-10-09 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest, NMB, Neuromuscular Blockade, Rocuronium
MeSH Terms: conditions — Heart Arrest | interventions — Rocuronium; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rocuronium (Experimental): Patients will receive a bolus dose of 1 mg/kg, then a continuous intravenous (IV) infusion as per standard intensive care unit practice.
  Of note, protocol allows for use of cistatracurium in place of rocuronium for either reasons of drug-shortage or clinical conditions (if institutional preferences for dose adjustment in liver or renal insufficiency arise).
  Interventions: Drug: Rocuronium
- Usual Care (Placebo Comparator): Patients will receive 100 mL of normal saline over 5-10 minutes at the beginning of the study in addition to usual care.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Rocuronium — Neuromuscular Blockade
  Arms: Rocuronium
Drug: Normal Saline — Normal Saline
  Arms: Usual Care

SUMMARY:
The main purpose of this study is to evaluate if neuromuscular blockade improves lactate clearance (and preliminary secondary clinical outcome measures) as compared to usual care in post-cardiac arrest patients undergoing targeted temperature management.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) occurs in more than 300,000 patients in the United States each year with an estimated mortality of greater than 90%. Unfortunately, we currently have little to offer in terms of treatment other than supportive care for the post-cardiac arrest patient. Neuromuscular blockade (NMB) is sometimes utilized in post-arrest patients particularly for the prevention of shivering. However, usage of NMB remains controversial and current American Heart Association (AHA) recommendations are to minimize utilization. Recent prospective randomized trials in patients with acute respiratory distress syndrome suggest a mortality benefit from NMB and an excellent safety profile. Furthermore, observational trials in both sepsis and post-cardiac arrest show that the use of NMB is associated with improved survival. Given this, we hypothesize that continuous NMB will be beneficial in post-arrest patients. In order to test this hypothesis, we propose a multi-center, randomized, open-label, phase II trial in post-CA patients comparing sustained NMB administration for 24 hours to standard of care after return of spontaenous circulation (ROSC). We will enroll adult, comatose OHCA patients with ROSC and will utilize an already existing clinical trials network for the completion of the study. Patients will be randomized to receive either rocuronium for 24 hours or to receive placebo with usual care. Previous data from our group has suggested that lactate levels in the post-arrest patient are a good surrogate marker for mortality. We have therefore chosen to utilize lactate levels at 24 hours as the primary endpoint for the current trial. Secondarily we will evaluate clinical endpoints including length of stay (LOS), in-hospital mortality, and good neurological outcome. We will perform a sub-study of inflammatory markers and oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Cardiac arrest with sustained return of spontaneous circulation (ROSC)
* Comatose (i.e., not following commands) following ROSC
* Undergoing targeted temperature management (TTM)
* Time of enrollment ≤ 6 hours from initiation of targeted temperature management
* Serum Lactate ≥2

Exclusion Criteria:

* Pre-existing dementia, severe brain injury, or dependence on others for activities of daily living (i.e. a modified Rankin scale (mRS) score of 4 or higher)
* Traumatic etiology of the cardiac arrest
* Protected population (pregnant, prisoner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-10; Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - Michael Kurz, Birmingham, Alabama
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Robert Swor, Royal Oak, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moskowitz A, Andersen LW, Rittenberger JC, Swor R, Seethala RR, Kurz MC, Berg KM, Chase M, Cocchi MN, Grossestreuer AV, Liu X, Holmberg MJ, Callaway CW, Donnino MW. Continuous Neuromuscular Blockade Following Successful Resuscitation From Cardiac Arrest: A Randomized Trial. J Am Heart Assoc. 2020 Sep;9(17):e017171. doi: 10.1161/JAHA.120.017171. Epub 2020 Aug 27. PMID 32851921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2014 and May 2019, we recruited adult patients (aged ≥18 years) who experienced a cardiac arrest and subsequently had sustained ROSC (≥20 minutes) but remained unresponsive and were undergoing TTM between 32℃ and 36℃. We added an additional inclusion criterion of a minimum serum lactate level of ≥2mmol/L early in study enrollment.
Pre-assignment Details: Of 818 patients assessed for eligibility, 83 met inclusion criteria and were randomized to treatment.
Groups:
- Rocuronium: Patients will receive a bolus dose of 1 mg/kg, then a continuous I.V. infusion as per standard intensive care unit practice.
  Of note, protocol allows for use of cistatracurium in place of rocuronium for either reasons of drug-shortage or clinical conditions (if institutional preferences for dose adjustment in liver or renal insufficiency arise).
  Rocuronium: Neuromuscular Blockade
Period: Overall Study
Arm/Group | Rocuronium | Usual Care
Started | 39 | 44
Completed | 37 | 43
Not Completed | 2 | 1
Not completed — 2 patients in NMB arm and 1 in control arm had clinical changes that precluded drug administration | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocuronium | Usual Care | Total
Number analyzed (Participants) | 37 | 43 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [57 to 77] | 64 [56 to 77] | 65 [56 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 20 | 29 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (n, % White) | 20 | 22 | 42
  Race (n, % Black/African-American) | 7 | 12 | 19
  Race (n, % Asian) | 1 | 0 | 1
  Race (n, % American Indian/Native Alaskan) | 1 | 0 | 1
  Race (n, % Other) | 2 | 0 | 2
  Race (n, % Unknown/Not Reported) | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 37 | 43 | 80
Past Medical History: Congestive Heart Failure [Count of Participants; unit: Participants] | 9 | 12 | 21
Past Medical History: Atrial Fibrillation [Count of Participants; unit: Participants] | 7 | 9 | 16
Past Medical History: Coronary Artery Disease [Count of Participants; unit: Participants] | 14 | 9 | 23
Past Medical History: Prior Cardiac Arrest [Count of Participants; unit: Participants] | 0 | 0 | 0
Past Medical History: Chronic Pulmonary Disease [Count of Participants; unit: Participants] | 12 | 9 | 21
Past Medical History: Liver Cirrhosis [Count of Participants; unit: Participants] | 1 | 2 | 3
Past Medical History: Kidney Disease [Count of Participants; unit: Participants] | 9 | 14 | 23
Past Medical History: Active Malignancy [Count of Participants; unit: Participants] | 3 | 2 | 5
Arrest Characteristics: Location (n, % Out of Hospital Cardiac Arrest) [Count of Participants; unit: Participants] | 35 | 40 | 75
Arrest Characteristics: Initial Rhythm (n, % Shockable) [Count of Participants; unit: Participants] | 17 | 16 | 33
Arrest Characteristics: Estimated Low-Flow Time (minutes, median, IQR) [Median (Inter-Quartile Range); unit: minutes] | 4 [0 to 7] | 2 [0 to 10] | 3 [0 to 10]
Arrest Characteristics: Witnessed (n, % yes) [Count of Participants; unit: Participants] | 27 | 26 | 53
Arrest Characteristics: Bystander Cardipulmonary Resuscitation (CPR) Provided (n, % yes) [Count of Participants; unit: Participants] | 24 | 26 | 50
Arrest Characteristics: Arrest Etiology (n, % cardiac) [Count of Participants; unit: Participants] | 27 | 30 | 57
Characteristics at Enrollment: Time from ROSC to Study Drug (hours, median, IQR) [Median (Inter-Quartile Range); unit: hours] | 7.5 [6 to 8.3] | 6.3 [5 to 7.5] | 6.5 [5.2 to 7.9]
Characteristics at Enrollment: pH (median, IQR) [Median (Inter-Quartile Range); unit: pH] | 7.3 [7.2 to 7.3] | 7.3 [7.2 to 7.4] | 7.3 [7.2 to 7.4]
Characteristics at Enrollment: Partial Pressure of Carbon Dioxide (pCO2) median, IQR [Median (Inter-Quartile Range); unit: mmHg] | 41.5 [34.5 to 53.5] | 40.0 [33.5 to 48.5] | 41.5 [34 to 49.5]
Characteristics at Enrollment: Partial Pressure of Oxygen (pO2) median, IQR [Median (Inter-Quartile Range); unit: mmHg] | 100.0 [76.0 to 168.5] | 161.0 [83.0 to 245.0] | 132.5 [79.5 to 232]
Characteristics at Enrollment: Shock Stratification (n, % shock) [Count of Participants; unit: Participants] — Shock stratification (n, %) refers to the number and percent of patients in each arm who were on vasopressors at the time of enrollment and therefore were considered to be in shock.
  Participants | 19 | 21 | 40
Characteristics at Enrollment: S-T Elevation Myocardial Infarction (STEMI) present (n, % yes) [Count of Participants; unit: Participants] | 4 | 6 | 10
Characteristics at Enrollment: Target temperature (median, IQR) [Median (Inter-Quartile Range); unit: celsius] | 35 [33.5 to 36] | 34 [33.5 to 35.5] | 35 [33.5 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Change in Lactate Over 24 Hours
Description: Change in median serum lactate level between enrollment and 24-hours after the receipt of study drug. A negative number indicates that the lactate levels were lower at 24 hours compared to their level at receipt of study drug.
Time Frame: 24 hours
Measure: Number; unit: mmol/L
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
mmol/L | -2.2 | -2.3

2. Primary Outcome: Change in Lactate Over 24 Hours: Effect Estimate
Description: Interaction between allocated treatment and time: ratio of geometric mean differences over 24 hours in log lactate values between the two groups.
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: Ratio
Groups:
- Effect Estimate: Value of the interaction term between allocated treatment and time, which is presented as a ratio of geometric mean differences over 24 hours. Values above 1.0 favor the placebo arm.
Arm/Group | Effect Estimate
Number analyzed (Participants) | 80
Ratio | 1.3 [1.0 to 1.8]

3. Secondary Outcome: Time ROSC to Target Temperature
Description: Time from return of spontaneous circulation to target temperature
Time Frame: Duration of hospitalization, limit 180 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
Hours | 6.8 [5.3 to 9.4] | 8.3 [4.7 to 11.2]
Statistical Analysis 1: Comparison: Rocuronium vs Usual Care; Test type: Equivalence — Time variable log transformed and compared using linear regression controlling for shock stratification and site. Effect estimate represents geometric mean difference. Values above 1.0 favor longer duration in the NMB arm; p = 0.82, Regression, Linear — A priori threshold for significance 0.05; Geometric mean difference = 1, 95% CI 2-sided [0.7 to 1.4]

4. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Description: Length of stay in ICU
Time Frame: Length of Stay Truncated at 28 Days
Population: ICU survivors row include only the 14 patients in each arm who survived to ICU discharge (n=14 in each arm).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
days
  All patients | 6.0 [3.0 to 11.0] | 4.0 [3.0 to 7.0]
  ICU survivors: number analyzed (Participants) | 14 | 14
  ICU survivors | 9.0 [6.0 to 16.0] | 5.0 [4.0 to 12.0]
Statistical Analysis 1: Comparison: Rocuronium vs Usual Care; All patients analyzed (N = 37 in NMB and 43 in Usual Care); Test type: Equivalence — LOS truncated at 28 days and compared using negative binomial regression controlling for stratification and site. Effect estimates represent incidence rate ratios. The parameter estimate, p value and CI provided below are from the negative binomial regression carried out all patients (N = 37 in NMB and 43 in Usual Care); p = 0.09, Negative binomial regression; Incidence rate ratio = 1.4, 95% CI 2-sided [1.0 to 1.9]
Statistical Analysis 2: Comparison: Rocuronium vs Usual Care; ICU survivors alone analyzed (n = 14 in each arm); Test type: Equivalence — LOS truncated at 28 days and compared using negative binomial regression controlling for stratification and site. Effect estimates represent incidence rate ratios. The parameter estimate, p value and CI provided below are from the negative binomial regression carried out on ICU survivors alone (n = 14 in NMB and 14 in Control); p = 0.35, Negative binomial regression; Incidence rate ratio = 1.3, 95% CI 2-sided [0.8 to 2.0]

5. Secondary Outcome: Mechanical Ventilation Duration
Description: Mechanical Ventilation Duration in Hours
Time Frame: Duration of hospitalization, limit 180 days
Population: Includes all patients, and also patients surviving to discontinuation of mechanical ventilation (n=14 in each group). Two patients discharged from the hospital on mechanical ventilation have duration truncated at time of discharge and are considered survivors to extubation.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
Hours
  All patients | 102.0 [64.3 to 206.4] | 82.7 [47.4 to 160.7]
  Survivors to extubation | 126.3 [76.1 to 280.6] | 66.9 [55.6 to 172.7]
Statistical Analysis 1: Comparison: Rocuronium vs Usual Care; Anaysis for the full data (n= 37 in NMB and 43 in Control); Test type: Equivalence — Duration log transformed and compared using linear regression controlling for shock stratification and site. Includes all patients (n=37 in NMB and n = 43 in control). Effect estimates represent geometric mean difference. Values above 1.0 favor longer duration in the NMB arm; p = 0.18, Regression, Linear; Duration log transformed and so parameter estimate represents geometric mean difference; Geometric mean difference = 1.3, 95% CI 2-sided [0.9 to 1.9]
Statistical Analysis 2: Comparison: Rocuronium vs Usual Care; Anaysis for the patients surviving to extubation (n= 14 in both groups); Test type: Equivalence — Duration log transformed and compared using linear regression controlling for shock stratification and site. Includes patients surviving to discontinuation of mechanical ventilation (n=14 in each group). Two patients discharged from the hospital on mechanical ventilation have duration truncated at time of discharge and are considered survivors to extubation. Effect estimates represent geometric mean difference. Values above 1.0 favor longer duration in the NMB arm; p = 0.32, Regression, Linear; Duration log transformed and so parameter estimate represents geometric mean difference; Geometric mean difference = 1.4, 95% CI 2-sided [0.7 to 2.9]

6. Secondary Outcome: Survival
Description: In-hospital survival
Time Frame: Duration of hospitalization, limit 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
Participants | 14 | 14
Statistical Analysis 1: Comparison: Rocuronium vs Usual Care; Test type: Equivalence — Comparison made using logistic regression controlling for shock stratification and site. Effect estimates represent odds ratios; p = 0.63, Regression, Logistic; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.5 to 3.3]

7. Secondary Outcome: Number of Participants With Rankin Score ≤3
Description: Modified Rankin scale to assess neurological outcome at discharge. The scale ranges from 0 to 6, and is used for measuring the performance of daily activities. The score is as follows:
  * 0: No symptoms
  * 1: No significant disability (able to carry out all usual activities, despite some symptoms)
  * 2: Slight disability (able to look after own affairs without assistance, but unable to carry out all previous activities)
  * 3: Moderate disability (requires some help, but able to walk unassisted)
  * 4: Moderately severe disability (unable to attend to own bodily needs without assistance, and unable to walk unassisted)
  * 5: Severe disability (requires constant nursing care and attention, bedridden, incontinent)
  * 6: Dead.
  Higher cores represent worse outcomes. Good and bad neurological outcome will be defined as a score of 0-3 and 4-6 respectively. This outcome reports the number of patients with a good neurological outcome( modified Rankin score ≤ 3)
Time Frame: Duration of hospitalization, limit 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
Participants | 11 | 9
Statistical Analysis 1: Comparison: Rocuronium vs Usual Care; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.35, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.6 to 4.7]

8. Secondary Outcome: Muscle Weakness Score
Description: Medical Research Council Scale : Measured for 6 muscle groups (3 in the upper limbs and 3 in the lower limbs). Maximum score is 30 (grade 5 for each group) and minimum is 0 (grade 0 for each group). If muscle group strength was not symmetric bilaterally, higher measurement used. Higher scores indicate better outcomes.
  Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3: Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed.
  Grade 2: Muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane.
  Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed
Time Frame: Duration of hospitalization, limit 180 days
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | Rocuronium | Usual Care
Number analyzed (Participants) | 37 | 43
Points | 30 [28 to 30] | 30 [27 to 30]

ADVERSE EVENTS:
Time Frame: From time of enrollment to time of discharge, an average of 7.2 days.
Arm/Group | Rocuronium | Usual Care
All-Cause Mortality (participants affected / at risk) | 23/37 | 29/43
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/43
Other Adverse Events (participants affected / at risk) | 0/37 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT02260258/SAP_000.pdf
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT02260258/Prot_001.pdf